CLINICAL TRIAL: NCT03884660
Title: Prospective Non-randomized Post Market Study Collecting Clinical Data on Safety and Effectiveness of the remedē® System
Brief Title: remedē System Therapy Study
Acronym: rēST
Status: Active, not recruiting | Type: Observational
Sponsor: Respicardia, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP1393
Record Dates: First submitted 2019-03-19; First posted 2019-03-21 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Central Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Central

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: remede System — Patients undergoing a remede System implant attempt. Study devices will be used per approved indications for use for each geography.

SUMMARY:
The purpose of this non-randomized post market study is to collect clinical data on the safety and effectiveness of the remedē System in a real-world setting.

DETAILED DESCRIPTION:
This is a multi-center, prospective, open label, non-randomized study to collect safety and effectiveness data in subjects with central sleep apnea implanted with the remedē System. Approximately 225 subjects will be enrolled and implanted at approximately 50 sites in the United States and Europe. A sub-study involving the WatchPAT device will be performed in a subset of sites.

ELIGIBILITY:
1. Moderate to severe central sleep apnea (AHI ≥ 15 events per hour) based on a sleep study scored by a local sleep laboratory. It is strongly recommended that a patient have a diagnostic PSG within 12 months of the expected implant date documenting moderate to severe CSA.
2. Age 18 years or older
3. Signed Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved informed consent
4. In the opinion of the investigator, subject is willing and able to comply with the protocol.
5. Not currently enrolled in another investigational study or registry that would directly interfere with the current study, except if the subject is participating in a mandatory government registry, or a purely observational registry with no associated treatments. Each instance should be brought to the attention of the sponsor to determine eligibility.
6. In the opinion of the Investigator, life expectancy exceeds one year.
7. The subject is not pregnant or planning to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are determined to be candidates, independent of this research study, to receive a de novo commercial implant of the remedē System are eligible for inclusion in this trial, subject to the entry criteria.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2019-06-18 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate safety of the remedē System at implant and protocol required follow up by assessment of serious adverse events (SAEs) related to procedure, device, or delivered therapy | 5 years
  Proportion of subjects with peri-operative and long-term serious adverse events (SAEs) related to the remedē System implant procedure, device or delivered therapy
Evaluate changes in sleep disordered breathing metrics after 12 months of therapy | 12 months
  Change from baseline to 12-month visit for the following sleep metrics measured during in-lab polysomnogram (PSG): apnea hypopnea index (AHI), central apnea index (CAI), oxygen desaturation index 4% (ODI4) and percent of sleep with oxygen saturation <90%

SECONDARY OUTCOMES:
Evaluate safety of the remedē System by assessment of non-serious AE related to procedure, device or delivered therapy | 5 years
  Proportion of subjects with non-serious AEs related to the remedē System implant procedure, device or delivered therapy
Evaluate changes in sleep disordered breathing metrics after 36 and 60 months of therapy | 36 and 60 months
  Change from baseline to 36- and 60-month visits for the following sleep metrics during an at home sleep apnea test (HSAT): apnea hypopnea index (AHI), central apnea index (CAI), oxygen desaturation index 4% (ODI4), percent of sleep with oxygen saturation <90%

OTHER OUTCOMES:
Evaluate changes in daytime sleepiness through 12 months | 12 months
  Epworth Sleepiness Scale (ESS) change from baseline to 12-month visit
Evaluate changed in quality of life (QOL) through 12 months | 12 months
  Quality of life assessment including the following:
  * Kansas City Cardiomyopathy Questionnaire (KCCQ) change from baseline at 12 months (HF subgroup only)
  * PROMIS-29 questionnaire change from baseline at 12, months
  * Patient Global Assessment (PGA) at 12 months
Evaluate changes in left ventricular ejection fraction in the HF subgroup after 12 months of therapy | 12 months
  Change in left ventricular ejection fraction based on echocardiographic assessment in the HF subgroup from baseline to 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Kathy McPherson, Study Director — ZOLL Respicardia, Inc.
Locations (32):
- United States (29):
  - Banner University Medical Center, Phoenix, Arizona
  - Arizona Heart Rhythm Center, Phoenix, Arizona
  - HonorHealth, Scottsdale, Arizona
  - The University of California San Francisco, San Francisco, California
  - University of Colorado- Anschutz, Aurora, Colorado
  - University of Colorado Health, Fort Collins, Colorado
  - Central Florida Pulmonary Group, Orlando, Florida
  - Emory University Midtown Hospital, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Michigan Health West, Wyoming, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - St. Luke's Mid America Heart Institute, Kansas City, Missouri
  - The Valley Hospital, Paramus, New Jersey
  - New Mexico Heart Institute - Lovelace Medical Center, Albuquerque, New Mexico
  - Northwell Health, New Hyde Park, New York
  - New York Presbyterian Hospital-Weill Cornell Medicine, New York, New York
  - Novant Health - Charlotte, Charlotte, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - The Ohio State Wexner Medical Center, Columbus, Ohio
  - Ohio Sleep Medicine Institute, Dublin, Ohio
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Monument Health, Rapid City, South Dakota
  - Baylor Scott and White - Dallas, Dallas, Texas
  - West Virginia University, Morgantown, West Virginia
- Netherlands (3):
  - OLVG Amsterdam, Amsterdam
  - Amphia Longresearch, Breda
  - Medisch Spectrum Twente, Enschede

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goldberg LR, Fox H, Stellbrink C, Bozkurt B, Boehmer JP, Mora JI, Doshi R, Morgenthaler TI, Levy WC, Meyer TE, McKane SW, Germany R; remede System Therapy Study Group. Design of the remede System Therapy (reST) study: A prospective non-randomized post-market study collecting clinical data on safety and effectiveness of the remede system for the treatment of central sleep apnea. Sleep Med. 2022 Dec;100:238-243. doi: 10.1016/j.sleep.2022.08.026. Epub 2022 Sep 6. PMID 36116293